CLINICAL TRIAL: NCT05038254
Title: There Is No Place Like Home- A Pragmatic Effectiveness Trial of Technology-Enhanced Outpatient Symptom Management to Reduce Acute Care Visits Due to Chemotherapy-Related Adverse Events
Brief Title: Enhanced Outpatient Symptom Management to Reduce Acute Care Visits Due to Chemotherapy-Related Adverse Events
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-0702; NCI-2021-07464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0702 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-30; First posted 2021-09-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Metastatic Colon Carcinoma; Metastatic Esophageal Carcinoma; Metastatic Gastric Carcinoma; Metastatic Liver Carcinoma; Metastatic Malignant Digestive System Neoplasm; Metastatic Malignant Small Intestinal Neoplasm; Metastatic Malignant Thoracic Neoplasm; Metastatic Pancreatic Carcinoma; Metastatic Rectal Carcinoma; Pathologic Stage IV Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IV Small Intestinal, Esophageal, Colorectal, Mesenteric, and Peritoneal Gastrointestinal Stromal Tumor AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (standard of care) (Active Comparator): Patients receive standard of care consisting of oncology care provided via telemedicine.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (standard of care, remote monitoring) (Experimental): Patients receive standard of care consisting of oncology care provided via telemedicine. Patients also undergo remote monitoring.
  Interventions: Other: Best Practice; Procedure: Patient Monitoring; Other: Questionnaire Administration
- Arm III (standard of care, remote monitoring, biometrics) (Experimental): Patient receive standard of care consisting of oncology care provided via telemedicine. Patients also undergo remote monitoring and biometric monitoring.
  Interventions: Other: Best Practice; Procedure: Patient Monitoring; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care telemedicine
  Other Names: standard of care; standard therapy
Procedure: Patient Monitoring — Undergo remote monitoring
  Other Names: medical monitoring; monitor
  Arms: Arm II (standard of care, remote monitoring); Arm III (standard of care, remote monitoring, biometrics)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies if enhanced outpatient symptom management with telemedicine and remote monitoring can help reduce acute care visit due to chemotherapy-related adverse events. Receiving telemedicine and remote monitoring may help patients have better outcomes (such as fewer avoidable emergency room visits and hospitalizations, better quality of life, fewer symptoms, and fewer treatment delays) than patients who receive usual care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of remote patient monitoring (RPM) on improving clinical outcomes.

SECONDARY OBJECTIVE:

I. Evaluate the following patient-centered outcomes: treatment delays, health-related quality-of-life (HRQOL), patient activation, and family caregiver-experience.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care consisting of oncology care provided via telemedicine.

ARM II: Patients receive standard of care consisting of oncology care provided via telemedicine. Patients also undergo remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* English- and Spanish-fluent participants with thoracic and/or gastrointestinal cancers who are scheduled to initiate or continue outpatient chemotherapy at either MDACC (Texas Medical Center campus and any Houston-area location) or MDACC oncology clinic at Lyndon B Johnson (LBJ) hospital
* Their adult (≥18 years) patient-identified or self-identified primary caregivers (MDACC only)
* Participants on combination chemotherapy and immunotherapy or combination chemotherapy and biologic will also be eligible for inclusion.
* Participants may participate if they do not have a caregiver, or if their caregiver declines participation; however, caregivers of MDACC participants may participate only if the participant consents.

Exclusion Criteria:

* Participants who are receiving investigational new drug treatments or concurrently enrolled in a phase 1 clinical trial will be excluded due to the associated structured reporting and regulatory requirements.
* Participants with a requirement for inpatient infusion (i.e. CAR-T cell therapy), living in institutional settings (i.e. prison, nursing homes), with a history of dementia, physical disability or neurological deficits that prohibit ability to report symptom burden will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of acute care visits | Up to 3 months
  Defined as the proportion of unique oncology patients with emergency room visits or hospital admission over a 3-month period.

SECONDARY OUTCOMES:
Change in health-related quality of life (HRQOL) | Baseline to 6 months
  HRQOL will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) Profile-29 version 2.1.
Change in patient engagement | Baseline to 6 months
  Patient engagement will be evaluated with the 13-item Patient Activation Measure (PAM), which assesses knowledge, skill, and self-efficacy for self-management of health
Change in symptom management | Baseline to 6 months
  Daily symptoms will be measured using the Common Terminology Criteria for Adverse Events version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan W Huey, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Offodile AC 2nd, Delgado D, Lin YL, Geyen D, Miller CJ, Jain S, Finder JP, Shete S, Fossella FV, Overman MJ, Peterson SK. Integration of Remote Symptom and Biometric Monitoring Into the Care of Adult Patients With Cancer Receiving Chemotherapy-A Decentralized Feasibility Pilot Study. JCO Oncol Pract. 2023 Jun;19(6):e811-e821. doi: 10.1200/OP.22.00676. Epub 2023 Feb 23. PMID 36821818
- See also: MD Anderson Cancer Center — http://www.mdanderson.org